CLINICAL TRIAL: NCT04243616
Title: Cemiplimab in High-risk or Locally Advanced Luminal and Triple Negative Breast Cancer (CemiHALT )
Brief Title: Cemiplimab in High-risk or Locally Advanced Luminal and Triple Negative Breast Cancer
Acronym: CemiHALT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Lubna Chaudhary, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00037175
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Invasive Breast Cancer
MeSH Terms: interventions — cemiplimab; Paclitaxel; Albumin-Bound Paclitaxel; Carboplatin; Doxorubicin; liposomal doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Drug Treatment (Experimental): Cemiplimab, Paclitaxel, Carboplatin (not mandatory), Doxorubicin, Cyclophosphamide
  Interventions: Drug: Cemiplimab; Drug: Paclitaxel; Drug: Carboplatin (not mandatory); Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cemiplimab — 350 mg, IV, Day 1 of Cycle 1-2 (3-week cycle)
  Other Names: Libtayo
Drug: Paclitaxel — 80 mg/m^2, IV, Day 1,8 and 15 of Cycles 1-4 (3-week cycle)
  Other Names: Taxol; Abraxane
Drug: Carboplatin (not mandatory) — Area under curve (AUC)=6, IV, Day 1 of Cycles 1-4 of Paclitaxel cycles (3-week cycle)
  Other Names: Paraplatin
Drug: Doxorubicin — 60 g/m^2, IV, Day 1 of Cycles 1-4 of ddAC (2-week cycle)
  Other Names: Lipodox; Lipodox 50; Doxil
Drug: Cyclophosphamide — 600 g/m^2, IV, Day 1 of Cycles 1-4 of dose-dense Adriamycin (Doxorubicin) and Cyclophosphamide (ddAC) (2-week cycle)
  Other Names: cytophosphane; Cytoxan; Neosar

SUMMARY:
This is a single-arm, open-label, phase 2 study that will enroll 36 subjects, who have pathologically proven diagnosis of invasive breast cancer, clinical stage tumor 1-3 (cT1-T3), node 0-3 (cN0-N3), metastasis 0 (cM0), hormone receptor positive (HR+) (estrogen-receptor-positive (ER+) and/or progesterone-receptor-positive (PR+) human epidermal growth factor receptor 2 (HER2) negative or hormone receptor-negative (HR-) (estrogen-receptor-negative (ER-) and progesterone-receptor-negative (PR-) human epidermal growth factor receptor 2 (HER2) negative/triple-negative breast cancer.

DETAILED DESCRIPTION:
Hypothesis: The addition of cemiplimab (PD-1 inhibitor) to standard neoadjuvant chemotherapy in patients with locally advanced HR+ HER2 negative or triple-negative (TN) breast cancer having positive PD-L1 and/or PD-L2 tumor expression will be associated with an increase in pathologic complete response of at least 20%.

Primary Objectives:

Assess pathologic responses in patients treated with neoadjuvant chemotherapy and cemiplimab.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven diagnosis of invasive breast cancer, cT1-T3, cN0-N3, cM0, HR+ (ER+ and/or PR+) HER2 negative or HR- (ER- and PR-) HER2 negative/triple negative breast cancer.
2. Tumors with positive PD-L1 and/or PD-L1 protein expression. Positivity is defined as PD-L1 and/or PD-L2 expression of ≥ 1% of immune cells within the stroma or in cancer cells.
3. Estrogen and/or progesterone receptor positive tumor defined ≥1% positively staining cells by immunohistochemistry, according to the current American Society of Clinical Oncology (ASCO) / College of American Pathologists (CAP) guidelines.
4. HER2/neu must be negative by immunohistochemistry (IHC) defined as IHC 0 or 1+ or fluorescence in situ hybridization (FISH) or other ISH methods with a ratio of < 2 according to current ASCO (American Society of Clinical Oncology)/CAP guidelines.
5. Candidate for neoadjuvant chemotherapy due to their clinical stage or subtype of breast cancer as decided by the treating physician.
6. Breast imaging with mammogram and/or ultrasound and/or MRI is per standard of care for diagnosis, but at least one modality of imaging must be completed within 30 days of registration.
7. Systemic imaging with CT scan, bone scan, positron emission tomography (PET) scan or MRI if clinically indicated per treating physician's discretion.
8. Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (per institutional normal) determined by echocardiogram or nuclear medicine scan within 30 days of registration.
9. The patient must be female.
10. Age ≥18 years.
11. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
12. The patient must provide study-specific informed consent prior to study entry.
13. Patients with a prior history of contralateral breast cancer will be considered eligible, if they have completed all treatment (including endocrine therapy) more than two years prior to registration.
14. Patients must not have had a prior treatment for this breast cancer or for any malignancy diagnosed or treated within the past two years, with the exception of non-melanomatous skin cancer, carcinoma in situ of the cervix and contralateral breast cancer, as described above.
15. Patients with bilateral breast cancer are also eligible provided HER2 negativity is documented on both right and left breast cancer and patient is deemed to be a candidate for neoadjuvant chemotherapy by treating physician.
16. Patients with multicentric or multifocal disease are eligible if they are a candidate for neoadjuvant chemotherapy.
17. Patients must meet one of the following:

    * Postmenopausal for at least one year before the screening visit, or
    * Surgically sterile, or
    * If they are of childbearing potential, negative pregnancy test within 14 calendar days prior to registration for women of childbearing potential
    * Women of childbearing age must use at least two adequate methods of contraception during the treatment period and at least 6 months from the last dose of chemotherapy. Examples of contraceptives include barrier methods, intrauterine devices (IUDs) hormonal or copper, oral contraceptive pills, and abstinence. Hormonal methods are not to be used by patients with HR+ breast cancer.
18. Adequate organ function with baseline lab values.

    * Absolute neutrophil count (ANC) ≥ 1500/µL
    * Hemoglobin (Hb) ≥ 8g/dL
    * Platelet count ≥ 100,000/µL
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3x institutional upper limit of normal (ULN)
    * Serum bilirubin within ≤ 1.5 x ULN except patients with Gilbert's syndrome for whom the direct bilirubin should be within normal range.
    * Creatinine clearance of ≥ 30 mL/min
    * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN. This applies to patients not receiving therapeutic anticoagulation. Patients on therapeutic anticoagulation should be on a stable dose.
    * Thyroid-stimulating hormone (TSH) ≤ institutional ULN

Exclusion Criteria:

1. Patients with clinical or pathologically proven metastatic disease.
2. HER2 positive disease as determined by either ISH or 3+ on IHC.
3. Synchronous non-breast malignancy (exceptions include non-melanomatous skin cancer, carcinoma in situ of the cervix).
4. Purely noninvasive breast cancer (i.e., ductal carcinoma in situ, lobular carcinoma in situ) without any concurrent invasive breast cancer
5. Men with breast cancer. Male breast cancer is a rare event.
6. Medical, psychiatric or other conditions that would prevent the patient from receiving the protocol therapy or providing informed consent.
7. Pregnant or lactating women are ineligible.
8. Treatment with any investigational drug within 30 days of registration. Prior treatment with any immunotherapy or chemotherapy for this breast cancer.
9. Current grade ≥ 2 peripheral neuropathy (according to NCI CTCAE v. 5.0).
10. Cardiopulmonary dysfunction defined as: Inadequately controlled angina, heart failure or serious cardiac arrhythmia not controlled by adequate medication.
11. Active Hepatitis B defined as positive Hep B surface antigen (HBsAg) or Hepatitis C. Patients with previous hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. If HBV DNA testing is positive, the patient is not eligible for study participation. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
12. Positive test for HIV.
13. History of symptomatic CHF⎯Grade ≥ 3 per NCI CTCAE v5.0 or New York Heart Association (NYHA) Class ≥ II.
14. History of autoimmune disease, including but not limited to myasthenia gravis, autoimmune myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

    * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
    * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible for this study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis) are eligible, provided the disease has no systemic manifestations and requires only low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%).
15. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (TNF) agents) within 2 weeks prior to study entry, or anticipated requirement for systemic immunosuppressive medications during the study. Patients who have received acute, low-dose, systemic immunosuppressant medications equivalent to ≤ 10mg of prednisone within the 7 days prior to study entry (small dose of dexamethasone for nausea, short course for upper respiratory tract infection etc.) may be enrolled in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2030-08-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with pathological complete response. | 27 weeks from start of treatment
  This is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lubna Chaudhary, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No